CLINICAL TRIAL: NCT05274802
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of ALS-4 (IM032) Administered Orally to Healthy Volunteers
Brief Title: A Study of ALS-4 in Healthy Adults Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptorum International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ALS-4-2020-11-01
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Healthy Subject

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part A1 (Single dose): Cohort A: ALS-4 25mg (Experimental): Single dose of ALS-4 or placebo before Breakfast
  Interventions: Drug: ALS-4; Drug: Placebo
- Part A1 (Single dose): Cohort B: ALS-4 50mg (Experimental): Single dose of ALS-4 or placebo before Breakfast
  Interventions: Drug: ALS-4; Drug: Placebo
- Part A1 (Single dose): Cohort C: ALS-4 100mg (Experimental): Single dose of ALS-4 or placebo before Breakfast
  Interventions: Drug: ALS-4; Drug: Placebo
- Part A1 (Single dose): Cohort D: ALS-4 200mg (Experimental): Single dose of ALS-4 or placebo before Breakfast
  Interventions: Drug: ALS-4; Drug: Placebo
- Part A1 (Single dose): Cohort E: ALS-4 300mg (Experimental): Single dose of ALS-4 or placebo before Breakfast
  Interventions: Drug: ALS-4; Drug: Placebo
- Part A2 (Single dose): Cohort F: ALS-4 50mg (Experimental): Dose three separate times in crossover fashion: (1) fasted morning dose; (2) fed morning dose; (3) fasted evening dose
  Interventions: Drug: Placebo; Drug: ALS-4
- Part B (Multiple dose): Cohort AA: ALS-4 50mg (Experimental): Multiple dose of ALS-4 or placebo up to two times daily
  Interventions: Drug: ALS-4; Drug: Placebo
- Part B (Multiple dose): Cohort BB: ALS-4 100mg (Experimental): Multiple dose of ALS-4 or placebo up to two times daily
  Interventions: Drug: ALS-4; Drug: Placebo
- Part B (Multiple dose): Cohort CC: ALS-4 200mg (Experimental): Multiple dose of ALS-4 or placebo up to two times daily
  Interventions: Drug: ALS-4; Drug: Placebo

INTERVENTIONS:
Drug: ALS-4 — Single dose of ALS-4 before Breakfast
  Other Names: IM032
  Arms: Part A1 (Single dose): Cohort A: ALS-4 25mg; Part A1 (Single dose): Cohort B: ALS-4 50mg; Part A1 (Single dose): Cohort C: ALS-4 100mg; Part A1 (Single dose): Cohort D: ALS-4 200mg; Part A1 (Single dose): Cohort E: ALS-4 300mg
Drug: Placebo — Single dose of placebo before Breakfast
  Arms: Part A1 (Single dose): Cohort A: ALS-4 25mg; Part A1 (Single dose): Cohort B: ALS-4 50mg; Part A1 (Single dose): Cohort C: ALS-4 100mg; Part A1 (Single dose): Cohort D: ALS-4 200mg; Part A1 (Single dose): Cohort E: ALS-4 300mg; Part A2 (Single dose): Cohort F: ALS-4 50mg
Drug: ALS-4 — Dose three separate times in crossover fashion: (1) fasted morning dose; (2) fed morning dose; (3) fasted evening dose
  Other Names: IM032
  Arms: Part A2 (Single dose): Cohort F: ALS-4 50mg
Drug: ALS-4 — Multiple dose of ALS-4 up to two times daily
  Other Names: IM032
  Arms: Part B (Multiple dose): Cohort AA: ALS-4 50mg; Part B (Multiple dose): Cohort BB: ALS-4 100mg; Part B (Multiple dose): Cohort CC: ALS-4 200mg
Drug: Placebo — Multiple dose of placebo up to two times daily
  Arms: Part B (Multiple dose): Cohort AA: ALS-4 50mg; Part B (Multiple dose): Cohort BB: ALS-4 100mg; Part B (Multiple dose): Cohort CC: ALS-4 200mg

SUMMARY:
A Phase I trial to evaluate the safety, tolerability and Pharmacokinetics of ALS-4 (IM032) in a single ascending dose (SAD) and multiple ascending dose (MAD) in healthy adult subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, first-in-human (FIH) study of ALS-4 (IM032) in healthy male and non-pregnant, non-lactating female volunteers. The study will consist of two phases: SAD and MAD. The study will evaluate the safety, tolerability and pharmacokinetic (PK) in 6 planned SAD cohorts (5 dose levels, and 1 cohort to evaluate for a potential food or circadian effect) with sentinel design (n=8 per cohort, total randomized 6 active: 2 placebo; sentinel design not applicable when a cohort with the same or a higher drug exposure has already been evaluated) and 3 planned MAD cohorts with sentinel design (n=8 per cohort, total randomized 6 active: 2 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male and female volunteers (18-60 years inclusive at the time of informed consent.)
* Body mass index (BMI) within 18.5 - 33.0 kg/m2 inclusive and weight >50 kg.
* Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
* QTc interval < 440 milliseconds for males and < 460 milliseconds for females, unless deemed otherwise by the PI/Sub-Investigator
* Systolic blood pressure between 95-140 mmHg, inclusive, and diastolic blood pressure between 55-90 mmHg, inclusive, and heart rate between 55-100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
* Clinical laboratory values within the most recent acceptable laboratory test range, and/or values are deemed by the PI/Sub-Investigator as "Not Clinically Significant".
* Ability to comprehend and be informed of the nature of the study, as assessed by staff. Capable of giving written informed consent prior to any study related procedure. Must be able to communicate effectively with clinic staff.
* Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
* Agree not to have a tattoo or body piercing until the end of the study.
* Subject agree to avoid pregnancy and use an acceptable highly effective method of contraception from at least 30 days prior to the study until at least 30 days after the last study procedure (IM032 or placebo).

Exclusion Criteria:

* Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first study drug administration, as determined by the PI/Sub-Investigator.
* Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.
* Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
* A known history or positive test result for human immunodeficiency virus (HIV), chronic Hepatitis B surface antigen, or Hepatitis C.
* A positive test result for drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), alcohol test and cotinine. Positive pregnancy test for female subjects.
* Known history or presence of Food allergies and/or presence of any dietary restrictions unless deemed by the - - PI/Sub-I as "Not Clinically Significant" or Severe allergic reactions
* Intolerance to and/or difficulty with blood sampling through venipuncture.
* Individuals who have donated, in the days prior to first study drug administration: 50-499 mL of blood in the previous 30 days; or 500 mL or more in the previous 56 days; or donation of plasma by plasmapheresis within 7 days prior to first study drug administration.
* Individuals who have participated in another clinical trial or who received an investigational drug within 30 days or 5-half-lives prior to first study drug administration.
* Use of any enzyme-modifying drugs and/or other products, including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (e.g., barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John´s Wort, and rifampicin) in the previous 30 days before first study drug administration.
* Use of any monoamine oxidase (MAO) inhibitors (e.g., phenelzine, tranylcypromine) within 30 days prior to first study drug administration.
* Use of any prescription medication within 14 days prior to first study drug administration (except for accepted methods of contraception).
* Use of any over-the-counter medications (including oral multivitamins, herbal and/or dietary supplements) within 14 days prior to first study drug administration (except for accepted methods of contraception).
* Consumption of food or beverages containing grapefruit and/or pomelo within 10 days prior to first study drug administration.
* Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing.
* Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by PI/Sub-Investigator.
* Have any other conditions that, in the opinion of the Investigator or Sponsor, would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study.
* Have had a tattoo or body piercing within 30 days prior to first study drug administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | Up to 28 days
  An adverse event is any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the Study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time-zero extrapolated to infinite time (AUCinf) | Up to 24 hours post dose
Area under the plasma concentration vs time curve from time 0 to the time of the last measurable concentration, or last sampling time t (AUCt) | Up to 24 hours post dose
Time of maximum observed plasma concentration (Cmax) | Up to 24 hours post dose
Time of maximum plasma concentration (Tmax) | Up to 24 hours post dose
Terminal elimination rate constant (λz) | Up to 24 hours post dose
Terminal elimination half-life(T1/2) | Up to 24 hours post dose
Plasma concentration at the end of the dosing interval at steady state on Day 14 (Ctau) | Up to 24 hours post dose
Minimum steady-state plasma concentration during a dosage interval on Day 14 (Cmin) | Up to 24 hours post dose
Maximum plasma concentration during a dosage interval (x = 1 or 14) (Cmax, Day x) | Up to 24 hours post dose
Area under the plasma concentration-time curve during a dosage interval on Day x (x = 1 or 14) (AUC12, Day x) | Up to 24 hours post dose
Accumulation ratio from Cmax from Day 1 to Day 14 (AR(Cmax)) | Up to 24 hours post dose
Accumulation ratio from AUC from Day 1 to Day 14 (AR(AUC)) | Up to 24 hours post dose
Time until maximum plasma concentration reached on Day x (x = 1 or 14) (Tmax,Day x) | Up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lee, PhD, Principal Investigator — Aptorum International Limited
Locations (1):
- BioPharma Services Inc., North York, Ontario, Canada